CLINICAL TRIAL: NCT06405854
Title: Effect of Coordination-based Exercise Intervention on Physical Fitness, Motor Competence and Executive Function in Preschool Children
Brief Title: Coordination-based Exercise Intervention in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Collaborators: Namik Kemal University (Other); Istanbul Aydın University (Other); Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Monira Aldhahi, Associate professor, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.198.10.22
Record Dates: First submitted 2024-05-04; First posted 2024-05-09 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Motor Skills; Balance; Fitness; Preschool
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: The participants, specifically the preschool children, may not be informed of their group assignment (Exercise Group or Control Group) to prevent behavior changes based on perceived expectations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coordination-based exercise intervention (Experimental): During the eight weeks, children in the coordinative exercise intervention group participated in sessions twice a week, each lasting 20 minutes. The foundational movement patterns tailored to the specific purpose were organized in a game format suitable for preschool-aged children. These foundational movement patterns comprise open-ended tasks progressing from simple to complex, with motor planning as a prerequisite. As the exercise intervention was game-based, the sessions were maintained as a fun, active, and social learning environment for the children.
  Interventions: Other: Exercise
- Control (No Intervention): The control group continued their regular preschool classes without any intervention.

INTERVENTIONS:
Other: Exercise — Children in the coordinative exercise intervention group will be encouraged to participate in sessions twice a week, each lasting 20 minutes. The foundational movement patterns tailored to the specific purpose were organized in a game format suitable for preschool-aged children. These foundational movement patterns comprise open-ended tasks progressing from simple to complex, with motor planning as a prerequisite. As the exercise intervention was game-based, the sessions were maintained as a fun, active, and social learning environment for the children. Duration of the intervention is eight weeks,
  Arms: Coordination-based exercise intervention

SUMMARY:
This study intended to assess the impact of coordination-based exercise interventions on physical fitness, motor competence, and executive function among preschoolers aged 4 to 6 years.

DETAILED DESCRIPTION:
Forty-four preschool children (22 boys and 22 girls), with a mean age of 5.90 years (SD = 0.28). Participants will be randomly assigned to an Exercise Group (n = 19) or a Control Group (n = 25). The Exercise Group will engage in 20-minute, fun, and game-based sessions focusing on foundational movement patterns appropriate for preschoolers, conducted twice weekly over eight weeks. In contrast, the Control Group continued with their regular unstructured school activities. Physical fitness was evaluated using agility tests, static-dynamic balance, and vertical jumping. Motor competence was assessed through the KTK3+ test battery, and inhibition control was measured using the Go/No-Go test. The study concluded that coordination-based exercises, structured around fun and engaging activities suitable for preschoolers, potentially enhance physical fitness, motor skills, and executive functions. These areas are essential for early childhood development, suggesting that integrating such exercises into preschool activities could be beneficial. However, specific results regarding the effectiveness of the interventions on the tested competencies would need to be detailed to confirm these hypothesized benefits fully. The study highlights the importance of structured physical activity in early childhood education settings for promoting essential developmental skills.

ELIGIBILITY:
Inclusion Criteria:

* typically preschoolers between the aged between 4-6 years old
* not taking any medication
* absence of cardiovascular, neurological, orthopedic, or psychiatric illnesses.

Exclusion Criteria:

• children with physical disabilities or other conditions that might significantly impact their ability to participate in the physical activity interventions might be excluded,

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Motor competence | at baseline and end of 8 week
  Motor competence will be assessed through the Body Coordination Test for Children (KTK). The Body Coordination Test for Children (KTK)+ test battery, supported by a hand-eye coordination task, will be used to assess the children's motor competence and it measures general gross motor coordination The Body Coordination Test for Children (KTK) test items include backward balancing (BB), sideways movement (MS), sideways jumping (JS), and hand-eye coordination tasks (EHC). All test items demonstrated good test-retest reliability: BB = 0.80, MS = 0.84, JS = 0.95, and EHC 0.87
Inhibition control (IC) | at baseline and end of 8 week
  IC will be measured using the Go/No-Go test. The Go/No-Go task is a protocol commonly used to measure inhibitory control in young children. The convergent validity of inhibitory control measurement has been observed to be good in this age group, with a strong correlation with the NIH Toolbox, which is frequently used and has a similar structure (r (80) = .40, p < 0.001). Additionally, internal consistency analyses of the Go/No-Go task revealed good reliability for the "Go" stimulus (Cronbach α = 0.95) and the "No-Go" stimulus (Cronbach 'sα = 0.84). In the Go/No-Go task, the children will be instructed to respond to the "go" stimulus (catch fish) by pressing the screen and to withhold their response to the "no-go" stimulus (avoid sharks). The practice trials consisted of 5 blocks of "catch fish" trials, five blocks of "avoid sharks" trials, and then a mixed block of 10 trials. After a short rest period, the task was completed with 75 stimulus trials divided into three test blocks (each
agility test | at baseline and end of 8 week
  The test course will be set with markers placed five yards (4.57m) to the left and right of the starting line, with indicators (motivational for the participants' age) placed accordingly. A photocell gate will be placed at the starting line to record repeated passage times. Before the start of the application, the participants took their position and when ready, they touched the marker on the right first, then the marker on the left, and finally crossed the starting line to complete the test.
Countermovement jump test | at baseline and end of 8 week
  Vertical jump performance was measured using an accelerometer (iVMES Athlete, Ankara, Turkey). During the test, the participants will be encouraged to jump as high as possible. The test was conducted twice with a 30-second rest between trials.

CONTACTS AND LOCATIONS:
Overall Officials: Monira I. Aldhahi, Principal Investigator — College of Health and Rehabilitation Sciences
Locations (1):
- Monira Aldhahi, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No